CLINICAL TRIAL: NCT02107313
Title: A Phase 1, Single Centre, Randomised, 2 Period Crossover Study to Determine the Effect of Food on the Pharmacokinetic Profile of a Single Dose of PBT2 Administered Orally to Healthy Volunteers
Brief Title: Phase 1 Study to Determine the Effects of Food on the Pharmacokinetic Profile of PBT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prana Biotechnology Limited (Industry)
Responsible Party: Sponsor
Organization: Pranabio (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PBT2-103
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fed Cohort (Other): PBT2 250 mg is administered orally following a high fat breakfast
  Interventions: Drug: Fed Cohort PBT2
- Fasted Cohort (Other): PBT2 250 mg is administered orally following a 10 hour period of fasting
  Interventions: Drug: Fasted Cohort PBT2

INTERVENTIONS:
Drug: Fed Cohort PBT2 — PBT2 250 mg is administered orally following a period of fasting for 10 hours and a high fat breakfast.
  Arms: Fed Cohort
Drug: Fasted Cohort PBT2 — PBT2 250 mg is administered orally after a period of fasting of 10 hours and without food
  Arms: Fasted Cohort

SUMMARY:
This study is designed to determine the pharmacokinetic (PK) profile of a single oral dose of PBT2 administered to healthy volunteers in the presence and absence of food.

DETAILED DESCRIPTION:
The study will be conducted in 2 dosing periods, with participants being randomised to receive PBT2 250 mg with or without food in the first dosing period, followed by a 7 day washout period before receiving the opposite fed/fasted condition to that allocated in the first dosing period. Pharmacokinetic samples will be collected during each dosing period, along with safety monitoring assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females with a BMI between 19 and 30kg/m2
* No clinically significant abnormalities

Exclusion Criteria:

* Exposure to medications/drugs that interfere with metabolism of PBT2 including drugs that inhibit or induce CYP1A2)
* Use of caffeine-containing beverages, supplements or alcohol within 72 hours of study entry
* Significant history of depression or other psychiatric illness
* Surgical or medical conditions which could significantly alter drug absorption, distribution, metabolism or excretion
* unable to swallow capsules

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Herd, Study Director — Prana Biotechnology
Locations (1):
- Centre for Clinical Studies - Nucleus Network, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at 1 site in Australia
Groups:
- Fed Cohort First Then Fasted Cohort: Per sequence, FED Cohort first then FASTED Cohort.
  Nine participants in the FED Cohort. PBT2 250 mg is administered orally following a high fat breakfast first, following a period of fasting for 10 hours and a high fat breakfast. Participants then cross over into the FASTED Cohort.
- Fasted Cohort First Then Fed Cohort: Per sequence, FASTED Cohort first, then FED Cohort.
  Nine participants in the Fasted Cohort. PBT2 250 mg is administered orally following a 10 hour period of fasting and without food first. Participants then cross over into the FED Cohort.
Period: Overall Study
Arm/Group | Fed Cohort First Then Fasted Cohort | Fasted Cohort First Then Fed Cohort
Started | 9 | 9 (One participant from the study did not cross over and participate in the FED cohort)
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — One participant did not do the FED cohor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants are first administered PBT2 250 mg orally following a period of fasting for 10 hours and a high fat breakfast in the FED cohort. Participants then cross over into the FASTED Cohort and receive PBT2 250 mg orally after a period of fasting of 10 hours and without food.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve (AUC 0-t)
Time Frame: prior to the initial doses on day 1 and 8 and then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8,10,12,16, 24, 30, 36, 48 hours post each dose
Population: PK Population, as defined as all participants who received at least one dose of PBT2 and had sufficient samples collected to determine PK parameters.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Fed Cohort: PBT2 250 mg is administered orally following a high fat breakfast
  Fed Cohort PBT2: PBT2 250 mg is administered orally following a period of fasting for 10 hours and a high fat breakfast. Participants cross over to the FASTED cohort after completing the Fed Cohort.
- Fasted Cohort: PBT2 250 mg is administered orally following a 10 hour period of fasting
  Fasted Cohort PBT2: PBT2 250 mg is administered orally after a period of fasting of 10 hours and without food. Participants cross over to the FED cohort after completing the Fasted Cohort.
Arm/Group | Fed Cohort | Fasted Cohort
Number analyzed (Participants) | 18 | 17
h*ng/mL | 1490.0 (542.0) | 1273.0 (552.3)

2. Secondary Outcome: Safety and Tolerability of PBT2 in Healthy Volunteers Measured by the Number of Participants Reporting at Least One Treatment Emergent Adverse Events
Time Frame: Up to 15 days after the first dose of PBT2
Population: Safety Population, as defined as all participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Fed Cohort | Fasted Cohort
Number analyzed (Participants) | 18 | 17
participants | 6 | 2

ADVERSE EVENTS:
Time Frame: All adverse events reported from time of consent to end of study (Day 15, which was 8 days since last dose of PBT2).
Arm/Group | Fed Cohort | Fasted Cohort
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 6/17 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fed Cohort (N=17) | Fasted Cohort (N=18)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less